CLINICAL TRIAL: NCT01781780
Title: Randomized Controlled Trial of Breakfast Recommendations on Weight: A Multi-Site Effectiveness Trial
Brief Title: Study of the Effectiveness of Breakfast Recommendations On Reducing Body Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Allison, Phd (Other)
Collaborators: University of Copenhagen (Other); University of Colorado, Denver (Other); Boston University (Other); Columbia University (Other)
Responsible Party: Sponsor-Investigator, David Allison, Phd, Professor, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: P30DK05633611
Record Dates: First submitted 2013-01-03; First posted 2013-02-01 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Obesity; Food Habits
Keywords: Obesity; Weight Loss; Breakfast
MeSH Terms: conditions — Obesity; Feeding Behavior; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- General Nutrition Recommendations (Active Comparator): Participants will be provided with a free USDA nutrition pamphlet describing general good nutrition habits. They will also receive an instruction handout to emphasize some of the points in the dietary guidelines in the handout. The clinician will go through both documents with participants in detail by reading them aloud and answering any questions, and it will be recommended that they incorporate the suggestions as best they can into their daily life.
  Interventions: Behavioral: General Nutrition Recommendations
- Breakfast Recommendation (Experimental): Participants randomized to the breakfast group will be instructed to consume breakfast before 10:00 a.m. every day, and will be asked to not eat again until after 11:00 a.m. Participants will be counseled on what a healthy breakfast is using an instruction handout. No specific restrictions will be given on types of foods that can be consumed for the breakfast meal. They will be instructed to keep track of their breakfast consumption (yes/no) using a calendar diary that will be provided to them. Participants will also be provided with a free USDA nutrition pamphlet describing general good nutrition habits. The clinician will go through both documents with participants in detail by reading them aloud and answering any questions, and it will be recommended that they incorporate the recommendations into their daily life as much as they can.
  Interventions: Behavioral: Breakfast Recommendation
- No Breakfast Recommendation (Experimental): Participants randomized to the no breakfast group will receive a detailed handout with instructions to not consume any calories before 11:00 a.m. every day. Only water or 0 calorie beverages may be consumed from the time of waking until 11:00 a.m. They will be instructed to keep track of their breakfast consumption (yes/no) using a calendar diary that will be provided to them. Participants will also provided with a free USDA nutrition pamphlet describing general good nutrition habits. The clinician will go through both documents with participants in detail by reading them aloud and answering any questions, and it will be recommended that they incorporate the recommendations into their daily life as much as they can.
  Interventions: Behavioral: No Breakfast Recommendation

INTERVENTIONS:
Behavioral: General Nutrition Recommendations
  Arms: General Nutrition Recommendations
Behavioral: Breakfast Recommendation
  Arms: Breakfast Recommendation
Behavioral: No Breakfast Recommendation
  Arms: No Breakfast Recommendation

SUMMARY:
This is an experiment that will compare the effect of recommending breakfast consumption, or breakfast skipping, on body weight. Our objective is to determine if breakfast consumption recommendations can produce weight loss, and if that weight loss is dependent on typical breakfast eating habits.

ELIGIBILITY:
Inclusion Criteria:

* Ages 20-65
* Men and women
* BMI ≥25, and ≤45 kg/m2
* Interested in weight loss
* Start day by 9:00 a.m. at least 5 days a week

Exclusion Criteria:

* Participation in any weight-reduction program, weight-loss diet, or other special diet within the previous 3 months.
* Weight loss or gain of >5% of body weight in the past 6 months for any reason except post-partum weight loss.
* Currently taking medication that suppresses or stimulates appetite.
* Currently regularly taking medication that requires eating with food in the morning as indicated on the prescription, or any non-steroidal anti-inflammatory drugs such as baby aspirin or Tylenol.
* History of prior surgical procedure for weight control or liposuction.
* Current smoker or quit smoking less than 6 months prior.
* Any major disease, including:

Active cancer or cancer requiring treatment in the past 2 years (except nonmelanoma skin cancer).

Active or chronic infections, including self-reported HIV positivity and active tuberculosis.

Active cardiovascular disease or event including hospitalization or therapeutic procedures for treatment of heart disease (e.g., coronary artery bypass, percutaneous transluminal coronary angioplasty) in the past 6 months; New York Heart Association Functional Class >2 with respect to congestive heart failure; stroke or transient ischemic attack in the past 6 months.

Gastrointestinal disease, including self-reported chronic hepatitis or cirrhosis, any episode of alcoholic hepatitis or alcoholic pancreatitis within past year, inflammatory bowel disease requiring treatment in the past year, recent or significant abdominal surgery (e.g., gastrectomy).

Active renal disease. Lung disease: chronic obstructive airway disease requiring use of oxygen. Diagnosed diabetes (type 1 or 2) and taking any anti-diabetic medications and/or controlling the disease via dietary manipulations.

Uncompensated or uncontrolled psychiatric disease (such as schizophrenia and bipolar disorder) that, in opinion of the investigators, would impede conduct of the trial or completion of procedures.

* A score on the Brief Symptom Inventory (BSI) (Derogatis & Melisaratos, 1983) that exceeds the 90th percentile.
* History of or current eating disorders, or an Eating Attitudes Test (EAT-26) score >20.
* Conditions or behaviors likely to effect the conduct of the trial: unable or unwilling to give informed consent; unable to communicate with the pertinent clinic staff; another household member is a participant or staff member in the trial; unwilling to accept treatment assignment by randomization; current or anticipated participation in another intervention research project that would interfere with the intervention offered in the trial; likely to move away from participating clinics before trial completed; unable to walk 0.25 mile in 10 minutes.
* Currently taking antidepressant, steroid, or thyroid medication, unless dosage has been stable for at least 6 months.
* A recent or ongoing problem with drug abuse or addiction.
* Excessive alcohol intake, either acute or chronic defined as any one of the following: 1) average consumption of 3 or more alcohol containing beverages daily; 2) consumption of 7 or more alcoholic beverages within a 24-hr period in the past 12 months; or 3) other evidence available to clinic staff.
* Willing to be randomized to any of the three experimental conditions.
* Pregnancy and childbearing: currently pregnant or less than 3 months post partum; currently nursing or within 6 weeks of having completed nursing; pregnancy anticipated during study; unwilling to report possible or confirmed pregnancies promptly during the course of the trial; unwilling to take adequate contraceptive measures if potentially fertile.
* Any other conditions which, in opinion of the investigators, would adversely affect the conduct of the trial.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Body Weight Change | Difference between baseline, and after 16 weeks
  Weight will be measured in light indoor clothes without shoes. Weight measurements will be recorded to the nearest 0.1 kg using a digital scale.

SECONDARY OUTCOMES:
Change in Body Mass Index | Difference between baseline and after 16 weeks
  BMI will be calculated as kg/m2.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Univeristy of Colorado Denver Anschutz Medical Campus, Denver, Colorado
  - Boston University, Boston Medical Center, Boston, Massachusetts
  - Columbia University, New York, New York
- Univeristy of Copenhagen, Copenhagen, Great Copenhagen, Denmark

REFERENCES:
- [Background] Schlundt DG, Hill JO, Sbrocco T, Pope-Cordle J, Sharp T. The role of breakfast in the treatment of obesity: a randomized clinical trial. Am J Clin Nutr. 1992 Mar;55(3):645-51. doi: 10.1093/ajcn/55.3.645. PMID 1550038
- [Derived] Dhurandhar EJ, Dawson J, Alcorn A, Larsen LH, Thomas EA, Cardel M, Bourland AC, Astrup A, St-Onge MP, Hill JO, Apovian CM, Shikany JM, Allison DB. The effectiveness of breakfast recommendations on weight loss: a randomized controlled trial. Am J Clin Nutr. 2014 Aug;100(2):507-13. doi: 10.3945/ajcn.114.089573. Epub 2014 Jun 4. PMID 24898236